CLINICAL TRIAL: NCT03501147
Title: The Effect of a Brief Daily Resistance Training Program in Healthcare Workers on Pain, Workability and Physical Function.
Brief Title: The Effect of a Resistance Training Program in Healthcare Workers on Pain, Workability and Physical Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, José Casaña Granell, Doctor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000260894
Record Dates: First submitted 2018-03-13; First posted 2018-04-18 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Musculoskeletal Pain; Physical Function; Work Ability
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 15 minutes of resistance training at the work place every day
  Interventions: Other: Resistance training
- Control (No Intervention): Usual work

INTERVENTIONS:
Other: Resistance training — 15 minutes of resistance training during work every day
  Arms: Intervention

SUMMARY:
The prevalence and consequences of musculoskeletal pain is considerable among healthcare workers, allegedly due to high physical work demands of healthcare work.

Performing physical exercise at the workplace together with colleagues may be more motivating for some employees and thus increase adherence. On the other hand, physical exercise performed during working hours at the workplace may be costly for the employers in terms of time spend. Thus, it seems relevant to perform a brief intervention. This study is intended to investigate the difference between the effect of workplace-based physical exercise (using elastic bands and body weight exercises) and a group control on musculoskeletal pain, physical exertion during work, physical function, need for recovery, self-rated use of analgesics, and work ability among healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare Workers at the Hospital
* Informed consent

Exclusion Criteria:

* Unable to perform exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Pain overall status: Standard 7-point patient global impression | 2 days after the end of intervention (POST)
  Standard 7-point patient global impression of pain collected at the endpoint

SECONDARY OUTCOMES:
Workability Index | Baseline
  Questionnaire work ability
Workability Index | 2 days after the end of intervention (POST)
  Questionnaire work ability
Physical function | Baseline
  Physical tests (push-ups, Biering-Sorensen test, Sit to Stand)
Physical function | 2 days after the end of intervention (POST)
  Physical tests (push-ups, Biering-Sorensen test, Sit to Stand)
Perceived physical exertion | Baseline
  Based on Borg's rate of perceived exertion (RPE) (Borg CR10 scale)
Perceived physical exertion | 3 weeks of resistance training
  Based on Borg's rate of perceived exertion (RPE) (Borg CR10 scale)
Perceived physical exertion | 6 weeks of resistance training
  Based on Borg's rate of perceived exertion (RPE) (Borg CR10 scale)
Perceived physical exertion | 2 days after the end of intervention (POST)
  Based on Borg's rate of perceived exertion (RPE) (Borg CR10 scale)
"Need for recovery scale" after work | Baseline
  Five point scale (1 = never, 5 = always)
"Need for recovery scale" after work | 3 weeks of resistance training
  Five point scale (1 = never, 5 = always)
"Need for recovery scale" after work | 6 weeks of resistance training
  Five point scale (1 = never, 5 = always)
"Need for recovery scale" after work | 2 days after the end of intervention (POST)
  Five point scale (1 = never, 5 = always)
Self-rated use of analgesics | Baseline
  The number of days the participants used analgesics during the last week
Self-rated use of analgesics | 3 weeks of resistance training
  The number of days the participants used analgesics during the last week
Self-rated use of analgesics | 6 weeks of resistance training
  The number of days the participants used analgesics during the last week
Self-rated use of analgesics | 2 days after the end of intervention (POST)
  The number of days the participants used analgesics during the last week
Pain: Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | Baseline
  Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10, 0 = not pain, 10 = worst possible pain)
Pain: Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | 3 weeks of resistance training
  Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10, 0 = not pain, 10 = worst possible pain)
Pain: Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | 6 weeks of resistance training
  Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10, 0 = not pain, 10 = worst possible pain)
Pain: Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10) | 2 days after the end of intervention (POST)
  Average pain intensity (Visual Analogue Scale (VAS) Scale 0-10, 0 = not pain, 10 = worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jose C Granell, PhD, Study Chair — University of Valencia
Locations (1):
- Clinic Universitary Hospital of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No